CLINICAL TRIAL: NCT03572127
Title: Does Obtaining the Majority of Dietary Protein From Non-animal Sources Support the Skeletal Muscle Adaptive Response to Structured Resistance Training in Young Men and Women
Brief Title: Mycoprotein, Resistance Training, and Hypertrophy
Acronym: HAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1718/27
Record Dates: First submitted 2018-05-21; First posted 2018-06-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophy
Keywords: Protein; Resistance Exercise; Skeletal Muscle; Mycoprotein; Sustainability
MeSH Terms: conditions — Hypertrophy | interventions — Diet

STUDY DESIGN:
Intervention Model Description: One group will consume a non-animal derived high protein diet, whilst the other group will consume a more traditional animal protein based diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-animal derived diet (Experimental): High protein diet derived from non-animal sources.
  Interventions: Other: Diet
- Animal derived diet (Active Comparator): High protein diet derived from animal sources.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — High protein diet derived from either animal or non-animal sources.

SUMMARY:
Protein is vital for the preservation of health and optimal adaptation to training. However, animal proteins come with economic and environmental issues. The study will investigate the effect of non-animal vs animal based habitual protein consumption on muscle protein metabolism and changes in muscle mass and function over a longer period of time.

DETAILED DESCRIPTION:
Protein is vital for the preservation of health and optimal adaptation to training. However, animal proteins come with a number of economic and environmental issues. Accordingly, the investigators need to develop an evidence base for more sustainable dietary proteins to support human nutrition. Mycoprotein is a non-animal protein produced by the continuous fermentation of the fungus Fusarium Venenatum. Previously, in a mechanistic study, it was determined that a single bolus of mycoprotein effectively supports muscle building in both rested and exercised skeletal muscle, to a similar extent as what would be expected of animal proteins. This suggests that similar adaptation of muscle tissue during training could be achieved when protein is obtained from non-animal derived protein sources.

The study will investigate the effect of high non-animal vs animal based habitual protein consumption on muscle protein metabolism and changes in muscle mass and function over a longer period of time. Initially, the study will employ a stable isotope tracer to quantify muscle protein synthesis over a period of three days in healthy male and female volunteers. During this time participants will consume a controlled vegan diet or an animal based diet, with daily unilateral resistance exercise. The second phase of the study will employ a 10 week diet and resistance training intervention, with the majority of a participant's protein either coming from animal or non-animal sources. This will determine the ability of a largely non-animal derived diet to support augmentations in muscle size and strength.

Briefly, participants will undergo 6 muscle biopsies over the course of an 11 week period. Initial biopsies will quantify muscle protein synthesis. Subsequent biopsies will characterise the adaptive response to the effects of nutrition and exercise. MRI scans will be employed to determine changes in muscle volume, and DXA scans will measure changes in body composition.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 40 years of age.
* Body mass index between 18 and 30.
* Recreationally active.
* Resistance training experienced (have previous performed resistance exercise, and are familiar with the basic movements).

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes) (as this may affect normal protein metabolism).
* Any diagnosed cardiovascular disease or hypertension (to avoid any complications associated with heavy exercise).
* Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥140mmHg over two or more measurements and an average diastolic blood pressure of ≥90mmHg over two or more measurements.)
* Chronic use of any prescribed or over the counter pharmaceuticals (that may modulate muscle protein metabolism).
* A personal or family history of epilepsy, seizures or schizophrenia.
* Allergic to mycoprotein / Quorn, penicillin, or milk.
* Pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 3 days
  Muscle protein synthesis measured via deuterium oxide

SECONDARY OUTCOMES:
Muscle fiber CSA | 10 weeks
  Changes in muscle fiber CSA
Muscle Strength | 10 weeks
  Changes in muscle strength
Muscle CSA | 10 weeks
  Changes in muscle CSA as measured by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Sports & Health Sciences, College of Life & Environmental Sciences, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Monteyne AJ, Coelho MOC, Murton AJ, Abdelrahman DR, Blackwell JR, Koscien CP, Knapp KM, Fulford J, Finnigan TJA, Dirks ML, Stephens FB, Wall BT. Vegan and Omnivorous High Protein Diets Support Comparable Daily Myofibrillar Protein Synthesis Rates and Skeletal Muscle Hypertrophy in Young Adults. J Nutr. 2023 Jun;153(6):1680-1695. doi: 10.1016/j.tjnut.2023.02.023. Epub 2023 Feb 22. PMID 36822394